CLINICAL TRIAL: NCT01317407
Title: Automatisierte Optische Überwachung Mittels Videosensorik Zur Verbesserung Der Patientensicherheit Auf Intensivstation (Automated Visual Monitoring for Improving Patient Safety (VIPSafe))
Brief Title: Automated Visual Monitoring for Improving Patient Safety (VIPSafe)
Acronym: VIPSafe
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Staedtisches Klinikum Karlsruhe (Other)
Collaborators: Karlsruhe Institute of Technology (Other)
Other Study IDs: SKKarlsruhe-VIPSafe
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Postoperative Confusion
Keywords: postoperative delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
After an operation many patients are in a confused mental status at the intensive care unit. In this status they possibly fall out of their bed or pull out endotracheal tubes or central venous catheters accidentally. For this, they need permanently monitoring and control through intensive care personnel.

The goal of the VIPSafe project is to develop robust techniques for automated patient monitoring, that rely on data from a small number of untethered sensors, which are nonetheless flexible enough to cope with a large variety of demands.

ELIGIBILITY:
Inclusion Criteria:

* patients with planned postoperative stay at intensive care unit after previous written consent to the study
* patients with not-planned postoperative stay at intensive care unit with written consent after admission to intensive care unit
* patients unfit to plead with admission to intensive care unit with written consent of the officially appointed agent

Exclusion Criteria:

* absent written consent
* age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a planned or not-planned stay at the intensive care unit after an operation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Anästhesie und Intensivmedizin, Städtisches Klinikum Karlsruhe, Karlsruhe, Germany